CLINICAL TRIAL: NCT07341152
Title: A Study to Assess the Pharmacokinetics and Relative Bioavailability of Crystalline LTG-001 Immediate Release Tablets Compared to LTG-001 SDD Formulation in Healthy Participants
Brief Title: A Study Comparing LTG-001 SDD Formulation To LTG-001 Crystalline Immediate Release Tablets In Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Latigo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LTG-001-011
Record Dates: First submitted 2025-12-02; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Period 1 Regimen A SDD Tablet (Experimental)
  Interventions: Drug: LTG-001 SDD
- Period 2 Regimen B (Experimental)
  Interventions: Drug: LTG-001 Formulation A Prototype 1
- Period 3 Regimen C (Experimental)
  Interventions: Drug: LTG-001 Formulation B Prototype 2
- Period 4 Regimen D (Experimental)
  Interventions: Drug: LTG-001 Formulation B prototype 2

INTERVENTIONS:
Drug: LTG-001 SDD — LTG-001
  Arms: Period 1 Regimen A SDD Tablet
Drug: LTG-001 Formulation A Prototype 1 — LTG-001
  Arms: Period 2 Regimen B
Drug: LTG-001 Formulation B Prototype 2 — LTG-001
  Arms: Period 3 Regimen C
Drug: LTG-001 Formulation B prototype 2 — LTG-001 High Dose
  Arms: Period 4 Regimen D

SUMMARY:
This is a single-center, open-label, part-randomized, crossover study in 14 healthy participants to assess the PK and safety profile of an SDD formulation of LTG-001 and two crystalline LTG-001 Instant Release tablet formulations, one of which will also be assessed at a differing dose level.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures.
* Must be willing and able to comply with all study requirements Aged 18 to 55 years inclusive at the time of signing informed consent.
* Must agree to use an adequate method of contraception (as defined in Section 9.4.
* Healthy males or non-pregnant, non-lactating, healthy females.
* Body mass index of 18.0 to 32.0 kg/m2 as measured at screening.
* Weight ≥50 kg at screening.

Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients.
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
* Significant serious skin disease, including rash, food allergy, eczema, psoriasis, or urticaria.
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease (except cholecystectomy), neurological or psychiatric disorder, as judged by the investigator.
* Have poor venous access that limits phlebotomy.
* Clinically significant abnormal clinical chemistry, hematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1). Participants with Gilbert's Syndrome are allowed.
* Has ALT or AST >1.5 × ULN; Total bilirubin >1.5 × ULN (for participants with known Gilbert's syndrome these criteria only apply if the total bilirubin >1.5 × ULN as long as direct bilirubin is ≤1.5 × ULN) at screening.
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <90 mL/min using the Cockcroft-Gault equation
* Positive HBsAg, HCV Ab or HIV antibody results at screening.
* Positive serum pregnancy test at screening or positive urine pregnancy test at first
* Participants who have received any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose. However, in no event shall the time between last receipt of IMP and first dose be less than 30 days.
* Participants who report to have previously received LTG-001. admission. Those who are pregnant or lactating will be excluded.
* Personal or family history of long QT syndrome or a QTcF interval > 450 msec for men or > 470 for women on screening or first admission ECG. Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g per day acetaminophen, HRT or oral contraception) in the 14 days before IMP administration (see Section 11.4). Exceptions may apply on a case-by-case basis, if considered not to interfere with the objectives of the study, as determined by the investigator.
* Participants who have had any vaccine within 15 days before first IMP administration History of any drug or alcohol abuse in the past 2 years.
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = 12 oz 1 bottle/can of beer, 1 oz 40% spirit, or 5 oz glass of wine).
* A confirmed positive alcohol urine test at screening or first admission.
* Current smokers and those who have smoked within the last 12 months.
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
* A confirmed positive urine cotinine test at screening or first admission.
* Positive drug screen test result at screening or first admission (drug of abuse tests are listed in Appendix 1) Donation of blood within 2 months or donation of plasma within 7 days prior to first dose of study medication.
* Participants who are, or are immediate family members of, a study site or sponsor employee.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-10-06 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Determine the relative bioavailability of two different LTG-001 crystalline formulations (test) compared to the LTG-001 SDD formulation (reference) in the fasted state. | From enrollment to Period 4, Day 3 Discharge
  results of LTG001 peak plasma concentration (Cmax)
Determine the relative bioavailability of two different LTG-001 crystalline formulations (test) compared to the LTG-001 SDD formulation (reference) in the fasted state | from enrollment to Period 4, Day 3 discharge
  Results of LTG001 Area under the plasma concentration versus time curve, (AUC (0-last))
Determine the relative bioavailability of two different LTG-001 crystalline formulations (test) compared to the LTG-001 SDD formulation (reference) in the fasted state. | from enrollment to Period 4, Day 3 discharge
  Results of LTG001 Area under the plasma concentration versus time curve, (AUC (0-inf))
To characterize the PK of LTG-001 and metabolites LTGO-4247 and LTGO-4449, following single administrations of up to two dose levels of two different LTG-001 IR tablet formulations in the fasted state. | From Enrollment to Period 4, Day 3 discharge
  Results of Cmax
To characterize the PK of LTG-001 and metabolites LTGO-4247 and LTGO-4449, following single administrations of up to two dose levels of two different LTG-001 IR tablet formulations in the fasted state | From enrollment to period 4, Day 3 Discharge
  Results of Tmax
To characterize the PK of LTG-001 and metabolites LTGO-4247 and LTGO-4449, following single administrations of up to two dose levels of two different LTG-001 IR tablet formulations in the fasted state. | enrollment to Period 4, Day 3 discharge
  Results of AUC(0-last)
To characterize the PK of LTG-001 and metabolites LTGO-4247 and LTGO-4449, following single administrations of up to two dose levels of two different LTG-001 IR tablet formulations in the fasted state. | from enrollment to Period 4, Day 3 discharge
  Results of AUC (0-inf)
To characterize the PK of LTG-001 and metabolites LTGO-4247 and LTGO-4449, following single administrations of up to two dose levels of two different LTG-001 IR tablet formulations in the fasted state. | from enrollment to Period 4, Day 3 discharge
  Results of T1/2

SECONDARY OUTCOMES:
Secondary Objective | from enrollment to Follow up phone call
  To assess safety and tolerability of single doses of LTG-001 when administered as IR formulations by evaluating number of participants with adverse events and SAEs, with abnormal laboratory tests results, abnormal 12-lead ECG readings, abnormal vital sign measurements and abnormal physical examination findings

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences - Miami, Inc, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No